CLINICAL TRIAL: NCT01538004
Title: Where Should Automated Blood Pressures be Done? RCT of BpTRU Measurement in Private or Non-private Areas of Primary Care Offices
Brief Title: Where Should Automated Blood Pressures be Done in Primary Care Offices?
Status: Withdrawn | Type: Observational
Why Stopped: Not funded
Sponsor: North Toronto Primary Care Research Network (Network)
Responsible Party: Principal Investigator, Michelle Greiver, Director of the North Toronto Primary Care Research Network, North Toronto Primary Care Research Network
Other Study IDs: 12-0217
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension
Keywords: Blood pressure determination; Primary health care; Office visits; Reproducibility of results
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BpTRU readings in private office area: Consenting patients will be randomly allocated using a random number table to BpTRU in an exam room. The first reading will be done with the research assistant present to ensure proper placement and recording and will then be left alone for the subsequent five measurements at one minute intervals. This will be immediately followed by a second set of readings in the alternate location. During both sets of readings the patient will be seated comfortably in a chair with arms and will be instructed not to talk or cross their legs. The same arm will be used for both sets of measurements with the blood pressure cuff at heart level. The average of the last five out of six blood pressure readings for each office location will be recorded. The decibel levels in each location will be recorded during BP readings using a Reed Sound Level Meter C-322. The patient's weight in kg, height in cm, gender and self reported history of hypertension will also be recorded.
- BpTRU readings in open office area: Consenting patients will be randomly allocated using a random number table to BpTRU in an open office area The first reading will be done with the research assistant present to ensure proper placement and recording and will then be left alone for the subsequent five measurements at one minute intervals. This will be immediately followed by a second set of readings in the alternate location. During both sets of readings the patient will be seated comfortably in a chair with arms and will be instructed not to talk or cross their legs. The same arm will be used for both sets of measurements with the blood pressure cuff at heart level. The average of the last five out of six blood pressure readings for each office location will be recorded. The decibel levels in each location will be recorded during BP readings using a Reed Sound Level Meter C-322. The patient's weight in kg, height in cm, gender and self reported history of hypertension will also be recorded.

SUMMARY:
The use of automated blood pressure measurement (ABPM) devices in the office setting is increasingly recognized as superior to manual BP measurement. Current guidelines recommend that patients be alone in a quiet room, with no interactions with health care professionals during the readings; in practice, this means using an exam room. However, we found no evidence supporting the location of ABPM. Furthermore, exam rooms are constantly being used in primary care offices, so this may not be practical in routine care.

For this study, fifty consecutive consenting patients age 18 or more in each of seven community based primary care offices will randomly be allocated to either ABPM in an exam room, or in a non-private area of the clinic. After being tested in the first location they will then be tested in the second location with the same device. The main outcome will be the mean value of the last five systolic blood pressures for each location within offices. Secondary measures will include blood pressures for patients with or without hypertension, a comparison of the initial and second set of blood pressures and of the effect of office noise in decibels on BP readings.

New technology is more readily adopted if barriers to use are minimized. If we find no differences in BP readings between office locations, clinicians will then have the option to use an additional office area to implement the automated BP measurement device.

DETAILED DESCRIPTION:
Following the design of our pilot study, patients consenting to two sets of blood pressure readings will be randomly allocated using a random number table to either automated blood pressure measurement using a BpTRU device in an exam room (private area without any traffic or staff) with the door closed, or BpTRU in an open (non-private area) of the clinic with routine office traffic and noise levels. Patients randomized to the private area first will be subsequently tested in the non-private area and those randomized to the non-private area first will then be tested in the private area. A single portable BpTRU machine will be used for all recordings. A research assistant will be trained on the use of the equipment with at least five supervised training readings. The BpTRU device will be placed on the patient's arm and readings will be recorded by the research assistant. The first reading will be done with the research assistant present to ensure proper placement and recording. The patient will then be left alone for the subsequent five measurements separated by one minute intervals. This will be immediately followed by a second set of readings in the alternate location. During both sets of readings the patient will be seated comfortably in a chair with arms and will be instructed not to talk or cross their legs. The same arm will be used for both sets of measurements with the blood pressure cuff at heart level. The research assistant will record the average of the last five out of six blood pressure readings for each office location, in accordance with the manufacturer's recommendations and previous studies.

The research assistant will record decibel levels in each location during BP readings using a Reed Sound Level Meter C-322 (Reed Instruments, Ste-Anne-de-Bellevue, Quebec, Canada). The sound level meter includes a data logger, and the mean decibel level per location for each set of readings will be recorded. The assistant will be trained in the use of the sound meter and logger and will use it during the five supervised BP training readings. The research assistant will also measure and record the patient's weight in kg, height in cm, and will collect information on patient's gender and self reported history of hypertension.

Planned sample size and analysis Our sample size is based on equivalence of BpTRU measurement done in non private office areas as compared to measurement done in private office areas, using the results of our pilot study. We consider differences of less than 5 mm Hg in systolic blood pressure to be clinically equivalent. In order to demonstrate equivalence for our primary outcome, and accounting for clustering effect in primary care offices, using a power of 80% and a two sided alpha level of 0.05 to conclude equivalency for a difference of 5 mm Hg or less, we will need to recruit 350 patients. Our planned recruitment is therefore fifty patients per office and seven office locations. 175 patients (25 per office location) will be randomly allocated to BpTRU measurement in a private exam room first and 175 will be allocated to an open area first.

Following the analytic methods used in our pilot study, we will use a random effect regression model to account for repeated measures within each participant for analyzing the data. Regression analysis will be undertaken to compare the measures and results will be adjusted for clustering effect. All tests will be two-sided using an alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age eighteen and over
* Able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive consenting patients age eighteen or over will be recruited from the waiting rooms of participating practices in Toronto, Ontario
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
mean value of the last five systolic blood pressures for each location within the offices | 1 hour
  comparison between the mean systolic values of the automated blood pressure measurements using a BpTRU device in private (quiet, no interactions with health care personnel) and non private areas of the offices.

SECONDARY OUTCOMES:
comparison of first and second sets of blood pressure readings | 1 hour
  Determination of rank effect on automated blood pressure measurements
comparisons of automated BP readings for patients with and without previously documented hypertension | 1 hour
effect of office decibel levels on automated office BP readings | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Greiver, MD MSc, Principal Investigator — North Toronto Primary Care Research Network
Locations (1):
- North Toronto Primary Care Research Network, Toronto, Ontario, Canada